CLINICAL TRIAL: NCT04396600
Title: The Professional Peer Resilience Initiative: Leveraging a Data-Driven Model to Maximize the Resilience of Healthcare Workers During the COVID-19 Pandemic
Brief Title: The Professional Peer Resilience Initiative
Acronym: PPRI
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: PSYCH-2020-28762
Record Dates: First submitted 2020-04-23; First posted 2020-05-20 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Stress; Stress Disorder; Stress, Psychological; Trauma, Psychological; Anxiety; Anxiety State; Post Traumatic Stress Disorder; Secondary Traumatic Stress; Professional Quality of Life; Stress Related Disorder; Stress Reaction; Stress Risk; Mental Resilience; Emotional Resilience
Keywords: Resilience; COVID-19; Coronavirus Disease 2019; Coronavirus; Healthcare Workers; Frontline; Traumatic Stress
MeSH Terms: conditions — Stress Disorders, Traumatic; Stress, Psychological; Psychological Trauma; Anxiety Disorders; Stress Disorders, Post-Traumatic; Compassion Fatigue; Fractures, Stress; COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthcare Workers Already Starting Peer Support Program
  Interventions: Behavioral: MinnRAP Peer Support Program
- Healthcare Workers Starting Peer Support Program Later
  Interventions: Behavioral: MinnRAP Peer Support Program

INTERVENTIONS:
Behavioral: MinnRAP Peer Support Program — The behavioral intervention consists of 1) pairing healthcare workers into "Battle Buddies" who maintain daily dialogue to detect stress and anxiety and 2) assigning a mental health consultant to each department to facilitate Battle Buddies and provide both small group sessions and individual psychological triage/referrals.

SUMMARY:
The Professional Peer Resilience Initiative (PPRI) study is an observational study aimed at understanding how symptoms of traumatic stress and resilience evolve over time in the University of Minnesota (UMN) healthcare workforce during the coronavirus disease 2019 (COVID-19) pandemic. The study is being conducted concurrently with a UMN peer support program called the MinnRAP program and will remotely administer quality of life and mental health surveys to healthcare workers before they start the MinnRAP program and throughout their participation in the program.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers (HCWs) and mental health consultants (MHCs) in UMN medical school departments

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of healthcare workers and mental health consultants in the University of Minnesota healthcare workforce.
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2024-11-10 (Actual)

PRIMARY OUTCOMES:
Change in professional quality of life | Before peer support program, through study completion (an average of 7 months)
  Professional Quality of Life Questionnaire (proQOL): min score of 10; max score of 50; higher scores mean worse outcome

SECONDARY OUTCOMES:
Change in mental health symptoms and resilience markers | Before peer support program, through study completion (an average of 7 months)
  Stress Risk & Resilience Self-Index: min score 0; max score of 12; higher scores mean worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Cristina S Albott, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States